CLINICAL TRIAL: NCT07003854
Title: Evaluation of the Effects of Mandibular Advancing Device in Obstructive Sleep Apnea Patients
Brief Title: Effects of Mandibular Advancing Device in Obstructive Sleep Apnea
Acronym: (MADs)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Serial 901
Record Dates: First submitted 2025-05-22; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: Mandibular advancing device
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Occlusal Splints

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- mild-moderate obstructive sleep apnea subjects (Experimental): receiving mandibular advancing devices
  Interventions: Device: Mandibular advancement device

INTERVENTIONS:
Device: Mandibular advancement device — Custom made titrable bi-bloc MADs worn during sleep to stabilize airway and treat obstructive sleep apnea

SUMMARY:
The goal of this clinical trial is to learn if Mandibular advancing devices work to treat obstructive sleep apnea in adults. Selected Participants have a mild or moderate degree of obstructive sleep apnea.The main questions it aims to answer are:

Do Mandibular advancing devices (MADs) lower the number of times participants experience apneas or hypopneas during sleep? Do MADs lower Apnea Hypopnea Index in adults when worn during sleep?

DETAILED DESCRIPTION:
This clinical trial aims to evaluate comprehensively the effects of a custom made titrable bi-block mandibular advancing device on the respiratory variables in polysomnography. This includes the apnea hypopnea index and the oxygen desaturation index. Also sleep variables such as sleep efficiency and snoring duration are evaluated. Also cone beam computed tomography scans are taken before treatment and after 6 weeks of using te appliance. the second CBCT scan is taken with the appliance intra-orally. The cahnge in airway volume and minimal axial area are measured.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years and older)
* Mild/Moderate obstructive sleep apnea
* Sufficient number of teeth( having at least one terminal molar)
* Healthy teeth and Periodontal ligament
* Good physical and mental capability helping the subjects to be able to deal with the appliance.

Exclusion Criteria:

* Severe OSA,
* Central sleep apnea,
* Pregnant females
* Somatic or psychological disease, or medications for psychological conditions.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
change in AHI | frpm enrollment to assessment of outcomes at least 8weeks
  difference between pre-tretment and post-treatment Apnea Hypopnea Index

CONTACTS AND LOCATIONS:
Overall Officials: Rania Mohamed Magdy, lecturer, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of dentistry AinShams University, Cairo, Abbaseya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Pre-treatment and post-treatment polsmnographic outcomes
Supporting Information: CSR
Time Frame: After one year of publication of results
Access Criteria: Anyone can access Polysomnographic data through personal communication

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/54/NCT07003854/Prot_SAP_000.pdf